CLINICAL TRIAL: NCT06774625
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study Evaluating the Efficacy and Safety of LTG 001 for Acute Pain After Surgical Removal of Impacted Third Molars
Brief Title: This is a Study Evaluating the Efficacy and Safety of LTG-001 for Acute Pain After Surgical Removal of Impacted Third Molars
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latigo Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LTG-001-003
Record Dates: First submitted 2024-12-23; First posted 2025-01-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain, Postoperative
Keywords: Acute Pain; Surgical Removal of Impacted Third Molars; Wisdom teeth
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LTG-001 High Dose (Experimental)
  Interventions: Drug: LTG-001 High Dose
- LTG-001 Mid Dose (Experimental)
  Interventions: Drug: LTG-001 Mid Dose
- LTG-001 Low Dose (Experimental)
  Interventions: Drug: LTG-001 Low Dose
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Suzetrigine (Active Comparator)
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: LTG-001 High Dose — LTG-001 High Dose
  Other Names: LTG-001
  Arms: LTG-001 High Dose
Drug: LTG-001 Mid Dose — LTG-001 Mid Dose
  Arms: LTG-001 Mid Dose
Drug: LTG-001 Low Dose — LTG-001 Low Dose
  Arms: LTG-001 Low Dose
Other: Placebo — Placebo
  Arms: Placebo
Drug: Suzetrigine — Active comparator - Nav1.8 inhibitor
  Arms: Suzetrigine

SUMMARY:
The goal of this clinical trial is to learn if LTG-001 works to treat pain after third molar removal surgery in adults. It will also learn about the safety of LTG-001. The main questions it aims to answer are:

Does drug LTG-001 treat the acute pain after surgical removal of impacted third molars (wisdom teeth) over 12 hours? How tolerable is LTG-001 after surgical removal of impacted third molars (wisdom teeth) over 12 hours?

Researchers in Part 1 will compare drug LTG-001 to a placebo (a look-alike substance that contains no drug) and in Part 2 to a placebo and a comparator to see if drug LTG-001 treats the post-surgical pain.

Participants will:

Take LTG-001 one time after the surgical removal of impacted third molars. Remain at the clinic for 12 hours after study dosing and return after a week for a safety check up.

Report the pain relief during the 12 hours after dosing to record changes in the post-operative pain

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged 18 to 50 years, inclusive, at the time of signing the informed consent
* Has a body weight ≥ 45 kg and a BMI ≤ 35 kg/m2.
* Subject requires extraction of 2 or more third molars, two of which must be mandibular molars that must be fully or partially bony, or combination of one fully and one partially bony impaction.
* Subject must agree to study required use of birth control.
* Post-surgical pain must meet protocol requirements.

Exclusion Criteria:

* Inability to take oral medications
* Prior dental surgery within 60 days or other surgical history that could confound surgery or post-operative procedures.
* History of impaired hepatic function or heart disease.
* Abnormal liver laboratories or other lab abnormality indicative of serious medical condition.
* Sensory abnormality that would confound post-surgery pain assessments.
* Chronic use of NSAIDs, benzodiazepines, opioid use within the last year, use of medications that prolong QTc intervals, or other dietary and medication restrictions.
* A subject with sleep apnea and/or on a home continuous positive airway pressure machine.
* Positive drug screen.
* Participant is under legal custodianship.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
SPID 0-12 | 12 hours
  Pain Intensity NRS Score change over the study.

SECONDARY OUTCOMES:
Perceptible Pain Relief | 12 hours
  Time to Confirmed Perceptible Pain Relief, assessed via 2-stopwatch technique.
Meaningful Pain Relief | 12 hours
  Time to Meaningful Pain Relief, assessed via 2-stopwatch technique.
Time to Rescue | 12 hours
  Time to first use of rescue medication.
TOTPAR over 0 to 12 hours | 12 hours
  Time-weighted summed pain relief as recorded on a sum of total pain relief (TOTPAR) over 0 to 12 hours (TOTPAR12) after the first dose of study drug.
2 Point Reduction in Pain on 0-10 Numerical Rating Scale | 12 hours
  Time to ≥ 2-point reduction in Numerical Rating Scale from baseline compared to placebo.
Global Evaluation | 12 hours
  Subject's global evaluation based on a 5-point scale asking, "Overall, how effective do you think the study drug is as a treatment for pain?"
No Required Rescue | 12 hours
  Subjects requiring no rescue opioid over 12 hours.
Total Rescue | 12 hours
  Total opioid rescue consumption over 12 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No